CLINICAL TRIAL: NCT04566471
Title: Palmoplantar Pustulosis and Generalized Pustular Psoriasis: A National Population-based Analysis of Prevalence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BI13680065
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-06

CONDITIONS: Palmoplantar Pustulosis; Generalized Pustular Psoriasis
Keywords: Generalized pustular psoriasis; Palmoplantar pustulosis; Urban Employee Basic Medical Insurance (UEBMI) data; prevalence; incidence
MeSH Terms: conditions — Psoriasis | interventions — Prevalence; Incidence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PPP and GPP: Palmoplantar pustulosis (PPP) and Generalized pustular psoriasis (GPP) are rare chronic inflammatory skin diseases, characterized by repeated episodes of sterile pustules in several months or years, associated with erythrokeratodermia generally. Both two diseases are easy to cause skin rupture, leading to bleeding and pain.
  Interventions: Other: prevalence/incidence

INTERVENTIONS:
Other: prevalence/incidence — It is an observational study for prevalence/incidence, no intervention provided.

SUMMARY:
This study plans to calculate the prevalence and incidence of palmoplantar pustulosis and generalized pustular psoriasis based on the national medical insurance data and analyze the composition characteristics and some clinical features of patients, through taking into account of the research status of palmoplantar pustulosis and generalized pustular psoriasis and the characteristics of medical insurance data.

ELIGIBILITY:
Inclusion Criteria:

* The insured population of the national urban employee basic medical insurance and the urban resident basic medical insurance from January 1, 2012, to December 31, 2016 (60 months) (the denominator)
* The patients have been diagnosed with palmoplantar pustulosis or generalized pustular psoriasis (including disease name, English abbreviation and ICD code)
* Both outpatient and inpatient patients are included

Exclusion Criteria:

* The individuals whose information is only contained in the reimbursement settlement database but not in the insurance coverage database will be considered as invalid reimbursement individuals and be excluded from the study (the denominator)
* The patients have been diagnosed with non-PPP and -GPP diseases, such as pustular psoriasis in palm and toe, pustular arthritis osteitis and SAPHO syndrome

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study used the Urban Employee Basic Medical Insurance (UEBMI) data from 2012 to 2016 to calculate the epidemiological characteristics of palmoplantar pustulosis and generalized pustular psoriasis. The database includes basic medical insurance data for urban workers and basic medical insurance data for urban residents, which covers 31 provinces, municipalities and autonomous regions. By the end of 2016, the number of people participating in the national basic medical insurance exceeded 1.3 billion, and the coverage rate of the insurance was stable at over 95%.
  The database is composed of an insurance coverage database and a reimbursement settlement database. The insurance coverage database involves demographic information, insurance information and payment information; and the reimbursement settlement database involves medical information, disease information and expense information.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of Palmoplantar pustulosis | From 2012 to 2016 in the Urban Employee Basic Medical Insurance (UEBMI) data of China
  Epidemiological characteristics of diseases: Mainly referring to indicators that could reflect the frequency related to the disease
prevalence of Generalized pustular psoriasis | From 2012 to 2016 in the Urban Employee Basic Medical Insurance (UEBMI) data of China
  Epidemiological characteristics of diseases: Mainly referring to indicators that could reflect the frequency related to the disease

SECONDARY OUTCOMES:
incidence of Palmoplantar pustulosis | From 2012 to 2016 in the Urban Employee Basic Medical Insurance (UEBMI) data of China
  Epidemiological characteristics of diseases: Mainly referring to indicators that could reflect the frequency related to the disease
incidence of Generalized pustular psoriasis | From 2012 to 2016 in the Urban Employee Basic Medical Insurance (UEBMI) data of China
  Epidemiological characteristics of diseases: Mainly referring to indicators that could reflect the frequency related to the disease
Economic burden of Palmoplantar pustulosis | From 2012 to 2016 in the Urban Employee Basic Medical Insurance (UEBMI) data of China
  Mainly referring to the consumption of medical resources, including medical expenses of patients.
Economic burden of Generalized pustular psoriasis | From 2012 to 2016 in the Urban Employee Basic Medical Insurance (UEBMI) data of China
  Mainly referring to the consumption of medical resources, including medical expenses of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Siyan Zhan, PhD, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No